CLINICAL TRIAL: NCT04830332
Title: Correlation of Preoperative Serum and Intraoperative Peritoneal Washing Fluid CA-125 Levels With Postoperative Tumor Histology in Patients With Endometrial Carcinoma: a Prospective-controlled Study
Brief Title: Correlation of Peritoneal Fluid CA-125 Levels With Postoperative Tumor Histology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erdemli State Hospital (Other)
Responsible Party: Principal Investigator, Suleyman Gunhan Doluoglu, Gynecologist, Erdemli State Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CA125
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Endometrial Carcinoma
Keywords: Endometrial carcinoma, CA-125, lymphovascular invasion
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Other): Women with endometrial carcinoma
  Interventions: Diagnostic Test: abdominal fluid CA-125 levels test

INTERVENTIONS:
Diagnostic Test: abdominal fluid CA-125 levels test — One hundred milliliters of normal saline was used as the abdominal washing liquid to obtain the sample for CA-125 measurement. Serum and abdominal washing fluid CA-125 levels were measured with a double antibody sandwich immunoenzymatic method, using Beckman Coulter DXI (Ireland) analyzer. I

SUMMARY:
In this prospective study, we aimed to investigate whether serum and abdominal washing fluid CA-125 levels correlated with postoperative histopathological parameters in patients with endometrial carcinoma.

DETAILED DESCRIPTION:
Endometrial cancer was diagnosed with histopathological examination of the samples obtained by dilatation and curettage. Preoperative serum CA-125 levels were determined in all patients. Serum and abdominal washing fluid CA-125 levels were measured with a double antibody sandwich immunoenzymatic method, using Beckman Coulter DXI (Ireland) analyzer. In addition to routine preoperative investigations, MRI was done in patients who were thought to have an extension outside the uterus.

During surgery, abdominal exploration was performed first, and then an abdominal fluid sample was obtained for cytological examination and measurement of CA-125 level. One hundred milliliters of normal saline was used as the abdominal washing liquid to obtain the sample for CA-125 measurement. Subsequently, total abdominal hysterectomy and bilateral salpingo-oophorectomy (TAH + BSO) were performed.

ELIGIBILITY:
Inclusion Criteria:

* Women with endometrial carcinoma

Exclusion Criteria:

* Previous history of any other malignancy
* Endometriosis
* Diagnosed with pelvic infection or with any other potential disease such as acute pancreatitis, colitis, diverticulitis, pericarditis, polyarteritis nodosa, Sjögren's syndrome and SLE

Ages: 55 Years to 68 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with endometrial carcinoma
Enrollment: 50 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2012-12-01 (Actual); Study Completion 2012-12-01 (Actual)

PRIMARY OUTCOMES:
Abdominal washing fluid CA-125 levels | One year

CONTACTS AND LOCATIONS:
Overall Officials: Suleyman G Doluoğlu, Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Reseacrh Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No